CLINICAL TRIAL: NCT01929291
Title: Assessment of Safety of GlaxoSmithKline (GSK) Biologicals' Combined Reduced Antigen Content Diphtheria-tetanus Toxoids and Acellular Pertussis Vaccine (dTPa), Boostrix When Administered According to the Approved Prescribing Information in Korea
Brief Title: Post-marketing Surveillance to Assess the Safety of Boostrix Vaccine Given According to Prescribing Information in Korea
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115374
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Diphtheria-Tetanus-acellular Pertussis Vaccines
Keywords: Korea; Post-marketing surveillance; Boostrix; Prescribing information; Safety
MeSH Terms: interventions — Boostrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Boostrix Group: Pre-adolescents (aged (≥10 years to ˂12 years), adolescents (aged ≥12 to ˂19 years), adults (aged 19 to 64 years) and elderly (≥ 65) who received Boostrix as a part of routine practice at a private clinic or hospital in Korea.
  Interventions: Biological: Boostrix; Other: Safety data collection

INTERVENTIONS:
Biological: Boostrix — Single intramuscular injection
  Other Names: dTPa vaccine
Other: Safety data collection — Safety monitoring: recording of adverse events using diary cards and recording of serious adverse events using the latest version of Korea's Post-Marketing Surveillance Serious Adverse Event Reporting Form

SUMMARY:
The purpose of this study is to collect safety information from pre-adolescents, adolescents and adults after Boostrix vaccination is administered according to the approved prescribing information in Korea.

DETAILED DESCRIPTION:
Protocol amendment 3 rationale was as follows:

* Age for analysis set is specified.
* Subjects with pregnancy will be analyzed by their pregnancy status before/after vaccination.
* Pregnancy notifications must be done within 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Written or signed informed consent obtained from the subject/ subject's parent(s)/Legally Acceptable Representative(s) of the child. Korean male or female subjects who were recently vaccinated or eligible to receive Boostrix according to the locally approved Prescribing Information.

Exclusion Criteria:

* Those who are not eligible for vaccination according to the local Prescribing Information.
* Child in care.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pre-adolescents, adolescents adults and elderly who receive Boostrix as a part of routine practice at a private clinic or hospital.
Sampling Method: Non-Probability Sample
Enrollment: 682 (Actual)
Dates: Start 2013-09-23 (Actual); Primary Completion 2016-01-11 (Actual); Study Completion 2016-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Suwon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park HJ, Kim SJ, Song R, Chen J, Kim JH, Devadiga R, Kang HC. A 6-year Prospective, Observational, Multi-Center Post-Marketing Surveillance of the Safety of Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis (Tdap) Vaccine in Korea. J Korean Med Sci. 2019 Mar 22;34(12):e105. doi: 10.3346/jkms.2019.34.e105. eCollection 2019 Apr 1. PMID 30940999

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 682 subjects case report forms were retrieved during the post-marketing surveillance period. Among those, 672 subjects were assessed for safety and the safety data from 10 subjects who did not fulfilled inclusion/exclusion criteria were analyzed separately.
Period: Overall Study
Arm/Group | Boostrix Group
Started | 672
Completed | 672
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Boostrix Group
Number analyzed (Participants) | 672
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.38 (14.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 451
  Male | 221
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 672

OUTCOME MEASURES:

1. Primary Outcome: Number of Unexpected Adverse Events (AEs)
Description: Unexpected AEs were defined as adverse events that are not reflected in the approved Prescribing Information in Korea.
Time Frame: During the 30-day (Day 0 - Day 29) follow-up period after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received the study vaccine.
Measure: Number; unit: Events
Arm/Group | Boostrix Group
Number analyzed (Participants) | 672
Events | 65

2. Primary Outcome: Number of Expected AEs.
Description: Expected AEs were defined as an adverse event that was expected from the subject during the post-vaccination follow-up period as described in the locally approved Prescribing Information in Korea.
Time Frame: During the 30-day (Day 0 - Day 29) follow-up period after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received the study vaccine.
Measure: Number; unit: Events
Arm/Group | Boostrix Group
Number analyzed (Participants) | 672
Events | 59

3. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or that was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the 30-day (Day 0 - Day 29) follow-up period after vaccination.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Boostrix Group
Number analyzed (Participants) | 672
Participants | 6

ADVERSE EVENTS:
Time Frame: AE(s) and SAE(s) were reported during the 6-Year Surveillance Period follow-up period after vaccination.
Arm/Group | Boostrix Group
All-Cause Mortality (participants affected / at risk) | 0/672
Serious Adverse Events (participants affected / at risk) | 6/672
Other Adverse Events (participants affected / at risk) | 90/672
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix Group (N=672)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Genital infection (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Birth premature (Reproductive system and breast disorders) | 1 (1)
Fever (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Boostrix Group (N=672)
Injection site pruritus (General disorders) | 3 (3)
Injection site rash (General disorders) | 2 (2)
Injection site anaesthesia (General disorders) | 1 (1)
Injection site warmth (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 14 (14)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux (Gastrointestinal disorders) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Common cold (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Labour premature (Reproductive system and breast disorders) | 4 (4)
Leukorrhoea (Reproductive system and breast disorders) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Birth premature (Reproductive system and breast disorders) | 1 (1)
Genital infection (Reproductive system and breast disorders) | 1 (1)
Pre-eclampsia (Reproductive system and breast disorders) | 1 (1)
Pruritus genital (Reproductive system and breast disorders) | 1 (1)
Vaginitis (Reproductive system and breast disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Skeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyuria (Renal and urinary disorders) | 2 (2)
Bacteriuria (Renal and urinary disorders) | 1 (1)
Cardiomegaly (Vascular disorders) | 1 (1)
Pressure blood increased (Vascular disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Foetal movements decreased (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Palpitation (Cardiac disorders) | 1 (1)
Injection site Pain (General disorders) | 21 (22)
Injection site Swelling (General disorders) | 5 (5)
Injection site Mass (General disorders) | 3 (3)
Injection site Erythema (General disorders) | 2 (2)
Injection site Tenderness (General disorders) | 2 (2)
Injection site Reaction (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Fever (General disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes